CLINICAL TRIAL: NCT00838968
Title: The Efficiency of Postoperative Interferon-alpha(IFNa) Treatment in p48 Positive Patients With Hepatocellular Carcinoma
Brief Title: The Efficiency of Postoperative Interferon-alpha Treatment in p48 Positive Patients With Hepatocellular Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we have found another marker (microRNA26) which is more sensitive to evaluate the effect of postoperative IFNa treatment in patients with HCC
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Liver cancer institute, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LCI
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; interferon-alpha; p48
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interferon-alpha; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interferon-alpha (IFN-alpha) (Active Comparator): the interferon-alpha is intramuscular injected 3,000,000U three times a week for 18 months
  Interventions: Drug: interferon-alpha
- control (No Intervention): no interventions were assigned

INTERVENTIONS:
Drug: interferon-alpha — interferon-alpha is intramuscularly or subcutaneously injected at 3,000,000-5,000,000 U three times a week for 18 months
  Other Names: Recombinant Human Interferon α1b for Injection; SINOGEN
  Arms: interferon-alpha (IFN-alpha)

SUMMARY:
The purpose of the study is to determine whether interferon-alpha is effective in the treatment of p48 Positive patients with HCC after curative resection.

DETAILED DESCRIPTION:
BACKGROUND: Postoperative interferon-alpha (IFN-alpha) therapy improved survival in patients with hepatocellular carcinoma (HCC). P48 is a predictive marker for outcome of postoperative interferon-alpha treatment in patients with HCC. Our study is to identify the Efficiency of Postoperative IFN-Alpha Treatment in p48 Positive Patients With HCC.

METHODS: An immunohistochemical study of P48 was performed on specimens that were collected from patients who underwent a curative resection of HCC. These patient with p48 Positive were randomized divided into a treatment group who received postoperative IFN-alpha therapy and a comparison group who not received. Besides the side effect, the overall survival rate and the disease-free survival rate will be observed.

Anticipated RESULTS: IFN alpha treatment improved the overall survival of p48 Positive patients with HCC after curative resection, probably by postponing recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with p48 Positive who underwent a curative resection of HCC

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
5-years survival rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hui-chuan Sun, MD, Principal Investigator — Liver Cancer Institute and Zhongshan Hospital, Fudan University, Shanghai, China